CLINICAL TRIAL: NCT03304834
Title: Minimally Invasive Treatment of Insufficient Superficial and Perforating Veins of the Lower Limb Using High Intensity Focused Ultrasound (HIFU): A Single Center Prospective Study
Brief Title: Treatment of Insufficient Superficial and Perforating Veins of the Lower Limb Using HIFU
Acronym: Archimedes01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theraclion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU-VV-001
Record Dates: First submitted 2017-10-03; First posted 2017-10-09 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Varicose Ulcer; Veins Diseases; Vein, Varicose
Keywords: HIFU; High intensity focused ultrasound
MeSH Terms: conditions — Varicose Ulcer; Varicose Veins | interventions — Compression Bandages

STUDY DESIGN:
Intervention Model Description: Monocentric study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ECHOPULSE (Experimental): Arm of patient treated by HIFU
  Interventions: Device: ECHOPULSE

INTERVENTIONS:
Device: ECHOPULSE — Patient are treated with the HIFU device and the physician is doing a compressive bandage.
  Other Names: Compression bandage

SUMMARY:
This is a single-center prospective study with a planned accrual of 35 patients with diagnosed symptomatic Lower Limb Veins System (Superficial, Perforating) Insufficiency (including recurrence at the thigh/groin level after previous treatment). The eligible patients must present a symptomatic Leg Veins System Insufficiency diagnosis which fulfills the inclusion/exclusion criteria. All patients will be consented at a Pre-Study Visit and evaluated for eligibility and for baseline characteristics of the disease. Patients will return to clinic on a separate day for the HIFU treatment. Device performance parameters will be collected during the HIFU visit. At follow-up visits at 3 days, 7 days and 3 months, changes in veins and flow characteristics will be evaluated by ultrasound and physical exam, and patient well-being, including pain and anxiety, will be evaluated by patient-reported VAS evaluations. Continued follow-up for a total of 3 months will be completed prior to subject study exit. Adverse events (AE) will be assessed at every study visit following HIFU treatment. An interim Safety Report will be issued after the first 5 patients will arrive at the 7 days visit and will be provided to the Ethics Committee. A second report will be issued once the first 5 patients will complete the follow-up period of 30 days and will be also provided to the Ethics Committee.

DETAILED DESCRIPTION:
The Echopulse System provides High Intensity Focused Ultrasound (HIFU) ablation of soft tissue. The energy is delivered via an extra-corporeal treatment probe, which includes an imaging system. The high-energy ultrasound waves propagate through the skin and are focused on a portion of the target tissue, generating intense heat and causing local cell apoptosis and progressive tissue volume reduction over the following months in the tissue within the focal area. The process is then repeated in a stepwise fashion to destroy the targeted tissues.

The Echopulse System is comprised of several components, including the console, treatment arm containing the visualization and treatment unit (VTU), and computer with touchscreen user interface. In addition, the Echopulse System is intended to be used in conjunction with a disposable cooling and coupling system known as EPack.

This is a single-center prospective study with a planned accrual of 35 patients with diagnosed symptomatic Lower Limb Veins System (Superficial, Perforating) Insufficiency (including recurrence at the thigh/groin level after previous treatment). The eligible patients must present a symptomatic Leg Veins System Insufficiency diagnosis which fulfills the inclusion/exclusion criteria. All patients will be consented at a Pre-Study Visit and evaluated for eligibility and for baseline characteristics of the disease. Patients will return to clinic on a separate day for the HIFU treatment. Device performance parameters will be collected during the HIFU visit. At follow-up visits at 3 days, 7 days and 3 months, changes in veins and flow characteristics will be evaluated by ultrasound and physical exam, and patient well-being, including pain and anxiety, will be evaluated by patient-reported VAS evaluations. Continued follow-up for a total of 3 months will be completed prior to subject study exit. Adverse events (AE) will be assessed at every study visit following HIFU treatment. An interim Safety Report will be issued after the first 5 patients will arrive at the 7 days visit and will be provided to the Ethics Committee. A second report will be issued once the first 5 patients will complete the follow-up period of 30 days and will be also provided to the Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for venous procedure involving lower limb superficial insufficiency, recurrence at the thigh/groin level or perforators incompetence.
* Physical condition allowing ambulation after the procedure.
* Availability of the patient for all the follow-up visits.
* Targeted tissue reachable for treatment with the device- meaning between 5mm and 26mm below the skin surface.
* Age over 18 years of age at the time of enrollment.
* No acute venous thrombosis.
* No complete, or near complete deep vein thrombosis.
* Patient has signed a written informed consent.

Exclusion Criteria:

* Patient is pregnant or nursing
* Known allergic reaction to anesthetics to be used
* Legally incapacitated or imprisoned patients
* Patient's vein target not clearly visible on the ultrasound images (in B mode) at the inclusion visit.
* Patient participating in another clinical trial involving an investigational drug, device or biologic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Reduction of venous reflux | 3 months
  as measured by ultrasound

SECONDARY OUTCOMES:
Measurement of flow abolition | 3 months
  As measured by ultrasound
Emergent Adverse Events | 3 months
  Measure of AEs and SAEs and adjunctive procedures for treating the reflux

CONTACTS AND LOCATIONS:
Overall Officials: Alfred OBERMAYER, MD, Principal Investigator — Karl Landsteiner Institut für funktionelle Phlebochirurgie
Locations (1):
- Karl Landsteiner Institut für funktionelle Phlebochirurgie, Melk, Austria

IPD SHARING:
Plan to Share IPD: No